CLINICAL TRIAL: NCT05189548
Title: To Evaluate the Safety and Primary Immunogenicity of Cell-free (Three-component) Combination Vaccine for Phase I Immunogenicity in Children and Infants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1004-F20210801
Record Dates: First submitted 2021-12-01; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-11

CONDITIONS: Safety、Immunogenicity
MeSH Terms: interventions — Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adsorbed a cell-free whitening break (three-component) combination vaccine (Experimental): A single-center and single-arm design was used to evaluate the safety and preliminary immunogenicity of the adsorbed cell-free leukiche (three-component) combination vaccine.
  Interventions: Biological: A single-center and single-arm design was used to evaluate the safety and preliminary immunogenicity of the adsorbed cell-free leukiche (three-component) combination vaccine

INTERVENTIONS:
Biological: A single-center and single-arm design was used to evaluate the safety and preliminary immunogenicity of the adsorbed cell-free leukiche (three-component) combination vaccine — A single-center and single-arm design was used to evaluate the safety and preliminary immunogenicity of the adsorbed cell-free leukiche (three-component) combination vaccine

SUMMARY:
A single-center and single-arm design was used to evaluate the safety and preliminary immunogenicity of the adsorbed cell-free leukiche (three-component) combination vaccine.Main purpose: To evaluate the safety of the adsorbed cell-free whitening break (three components) combination vaccine;Secondary purpose: To preliminarily evaluate the immunogenicity of the adsorbed cell-free whitening break (three components) combination vaccine.

DETAILED DESCRIPTION:
Main endpoint:

1. Adverse events within 30 minutes after vaccination of each test dose;
2. occurrence of solicitation adverse events within 0-7 days after vaccination of each dose;
3. The occurrence of non-solicitation adverse events within 0-30 days after vaccination for each test dose;
4. occurrence of serious adverse events 6 months after the first dose of immunization to the whole immunization.

Secondary endpoint:

1. Abnormal occurrence of laboratory test indicators on day 4 after immunization between 4 and 6 years old age groups;
2. Geometrical mean concentration (GMC) or geometric mean titer (GMT) of each antibody combined with the cell-free whitening break (three components) for 30 days after the full basal immunization in the 3-month age group;
3. Geometrical mean concentration (GMC) or geometric mean titer (GMT) of each antibody combined with cell-free leucocyte (three-component) adsorption at 30 days after 18 to 24 months of age immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent and healthy people aged 4-6 years old, 18-24 years old, and March age group (90-119 days);
2. Children between the ages of 4 and 6 who complete the whole immunization (4 doses) and do not receive diphtheria tetanus combination vaccine according to diphtheria and immunization program procedures;
3. Children of age groups from 18 to 24 who complete the basic immunization (3 doses) and do not strengthen the immunization according to the immunization planning program;
4. Infants of the age of March who were not vaccinated with one hundred whitening components, 13-valent pneumonia polysaccharide-binding vaccine and Hib vaccine;
5. Obtain the informed consent from the subject's legal guardian, and sign the informed consent form;
6. The legal guardian of the subject can comply with the requirements of the clinical trial protocol;
7. The axillary body temperature of the subject was 37.0℃.

Exclusion Criteria:

1. Ablaboratory examination indicators for children aged 4 to 6, except minor abnormalities judged by doctors without clinical significance;
2. A history of pertussis, diphtheria, and tetanus;
3. Infants born with preterm birth (birth before the 37th week of gestation), abnormal labor period (dystocia, instrumental midwifery, etc.), low weight (<2500g male and <2300g female); only at 3 months of age;
4. Innate malformations or developmental disorders, genetic defects, serious malnutrition, etc.;
5. Patients with epilepsy, convulsions or convulsions, or a family history of psychosis;
6. Autoimmune diseases or immune defects, or parents or siblings have autoimmune diseases or immune defects;
7. No splenic function and defective spleen function caused by any condition;
8. Abnormal coagulation function (such as lack of coagulation factors, abnormal coagulation disease, platelet), or obvious hematoma or coagulation disorder;
9. allergic to a known component of the study vaccine or any previous history of severe allergy (extensive urticaria, angioedema, etc.);
10. Immunoglobulin and / or any blood products (except hepatitis B immunoglobulin) were given within 3 months before the enrollment;
11. Those treated with any immunoenhancement or inhibitor within 3 months (continuous oral or infusion for more than 14 days;
12. Received subunit or inactivated vaccine in the past 7 days, and received live attenuated vaccine in the past 14 days;
13. Acute attacks of various acute diseases or chronic diseases in the past 7 days;
14. According to the investigator, the subject had any other factors not suitable to participate in the clinical trial.

The 2 and 3rd vaccination exclusion / delay criteria:

Exclusion criteria The investigator will terminate the subject vaccination trial vaccine if any of the following occurs.

1. Any newly diagnosed or suspected autoimmune disease or immunodeficiency disease issued during vaccination;
2. Other serious adverse events related to the study vaccine (including severe pain, severe swelling, severe limited restriction, persistent high fever, severe headache or other systemic or local reactions) occurred;
3. Severe allergic reaction or hypersensitivity reaction after vaccination (including severe urticaria / rash occurring within 30 minutes after vaccination);
4. The investigator evaluates any other reasons considered necessary to terminate the trial vaccination.

Delay the standard If any of the following conditions occur, the investigator will delay vaccination until the situation eases.The delay in vaccination should be kept within the specified time window (see: study flowchart).

1. Received subunit or inactivated vaccine in the past 7 days, and received live attenuated vaccine in the past 14 days;
2. At the time of vaccination, an acute disease (acute disease is a moderate or severe disease with or without fever) or a new chronic disease;
3. Physical examination of arm temperature> 37.0℃ before vaccination;
4. Other situations where the researchers believe that the vaccination should be postponed.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The safety of the adsorbed cell-free whitening break (three-component) combination vaccine was evaluated | Ten months
  1. Adverse events within 30 minutes after vaccination of each test dose;
  2. occurrence of solicitation adverse events within 0-7 days after vaccination of each dose;
  3. The occurrence of non-solicitation adverse events within 0-30 days after vaccination for each test dose;
  4. occurrence of serious adverse events 6 months after the first dose of immunization to the whole immunization.

SECONDARY OUTCOMES:
Immunimmunogenicity of the cell-free (three-component) combination vaccine was evaluated | Ten months
  1. Abnormal occurrence of laboratory test indicators on day 4 after immunization between 4 and 6 years old age groups;
  2. Geometrical mean concentration (GMC) or geometric mean titer (GMT) of each antibody combined with the cell-free whitening break (three components) for 30 days after the full basal immunization in the 3-month age group;
  3. Geometrical mean concentration (GMC) or geometric mean titer (GMT) of the cell-free leucocyte (three components) at 30 days after 18 to 24 months of age immunization.

CONTACTS AND LOCATIONS:
Locations (1):
- Santai County Center for Disease Control and Prevention, Mianyang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No